CLINICAL TRIAL: NCT00005961
Title: A Phase II Trial of O6-Benzylguanine (NSC 637037) and BCNU (Carmustine) in Patients With Metatstatic Melanoma
Brief Title: O6-benzylguanine and Carmustine in Treating Patients With Unresectable Locally Recurrent or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02340; UCCRC-10325; CWRU-1699; NCI-T99-0111; CDR0000067943 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2003-04

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — O(6)-benzylguanine; Carmustine

ARMS (1):
- Arm I (Experimental): Patients receive O6-benzylguanine IV over 1 hour, followed 1 hour later by carmustine IV over 1 hour on day 1. Treatment continues every 6 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: O6-benzylguanine; Drug: carmustine

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: carmustine

SUMMARY:
Phase II trial to study the effectiveness of O6-benzylguanine and carmustine in treating patients who have unresectable locally recurrent or metastatic melanoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than once chemotherapy drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective clinical response rate and duration of response in patients with unresectable locally recurrent or metastatic melanoma treated with O6-benzylguanine and carmustine.

II. Compare the toxicities of this regimen in patients with no prior chemotherapy vs prior chemotherapy failure.

III. Correlate clinical response to this regimen in these patients with O6-alkylguanine DNA alkyltransferase (AGT) depletion and baseline AGT in peripheral blood mononuclear cells and tumor tissue.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (chemotherapy failure vs chemotherapy naive).

Patients receive O6-benzylguanine IV over 1 hour, followed 1 hour later by carmustine IV over 1 hour on day 1. Treatment continues every 6 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.

Patients with disease progression are followed every 6 months. All other patients are followed every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven unresectable locally recurrent or metastatic melanoma

  * Chemotherapy naive with no more than 2 prior immunotherapy regimens (including cytokines, vaccines, or adjuvant interferon) OR
  * Prior chemotherapy failure with no more than 2 prior immunotherapy regimens (including adjuvant interferon) and no more than 1 prior chemotherapy regimen (which may include carmustine) not including antiangiogenesis therapy
* Measurable disease

  * At least 20 mm in at least 1 dimension by conventional technique OR at least 10 mm in at least 1 dimension by spiral CT scan
* No disease confined only to the CNS
* No uncontrolled symptomatic brain metastases regardless of other disease sites

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST and/or ALT no greater than 3 times upper limit of normal
* PT normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Pulmonary:

* DLCO at least 70% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent significant psychiatric or medical illness, including active infections, that would interfere with study therapy or increase risk
* No other malignancy within the past 5 years except curatively treated nonmelanomatous skin cancer, carcinoma in situ of the cervix, or superficial bladder cancer

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* At least 4 weeks since prior systemic chemotherapy (at least 6 weeks since prior carmustine or mitomycin) and recovered
* No other concurrent chemotherapy or investigational antineoplastic drugs

Radiotherapy:

* At least 2 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* At least 3 weeks since prior major surgery and recovered

Other:

* At least 4 weeks since other prior anticancer systemic therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-06; Primary Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Gajewski, MD, PhD, Study Chair — University of Chicago
Locations (13):
- United States (13):
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Mercy Ireland Cancer Center, Canton, Ohio
  - Ireland Cancer Center, Cleveland, Ohio